CLINICAL TRIAL: NCT06800690
Title: Role of Metabolic Sensing in Human Sweet Taste
Brief Title: Impact of Menstrual Phase on Oral Glucose Sensitivity
Status: Completed | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Paul A Breslin, Distinguished Professor, Rutgers, The State University of New Jersey
Other Study IDs: 2019001483; R21DC020365 (NIH)
Record Dates: First submitted 2025-01-17; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Ovulation; Menstruation
Keywords: estrogen; progesterone; glucose; sensitivity; taste; K-ATP
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cycling Women: This is a group of women who have regular menstrual cycles.
  Interventions: Diagnostic Test: Urinary Estrogen Level
- Men: These men serve as an age-matched control who do not have high estrogen levels, as males do not have menstrual cycles.
  Interventions: Diagnostic Test: Urinary Estrogen Level

INTERVENTIONS:
Diagnostic Test: Urinary Estrogen Level — Women had urinary estrogen metabolite levels measured daily to identify both the nadir (menstruation) and the peak (peri-ovulation) of the cycle. Men were also tested at the same time intervals, approximately two-weeks apart.

SUMMARY:
In this study we are determining whether the hormones associated with the phases of the menstrual cycle (menstruation & ovulation) influence taste sensitivity to glucose. We hypothesized that women would be more sensitive to oral glucose as assessed by absolute detection threshold during ovulation than when assessed during menstruation. These phases of the cycle are associated with peak plasma estradiol levels and nadir estradiol levels. There is evidence that estrogen can increase the sensitivity of the metabolic signaling pathway of the pancreatic beta-islet cells to stimulate insulin release more readily when glucose is present by increasing sensitivity of the K-ATP channel to ATP. Since the same metabolic signaling pathway is reported to be present in taste tissue, we tested whether peak estrogen levels would enhance taste detection of glucose but not sweeteners that cannot generate ATP, such as sucralose or methyl-D-glucopyranoside (MDG).

DETAILED DESCRIPTION:
Participants: The participants consisted of 15 healthy, non-obese, cycling females between the ages of 18-46 years. All participants completed informed consent and the study protocol was approved by the Rutgers University Institutional Review Board. 30 participants were screened for eligibility requirements. Inclusion criteria consisted of a regular menstrual cycle of 21-35 days. Exclusion criteria included hormonal contraceptives or other hormonal treatments, a history of polycystic ovarian syndrome (PCOS), menstrual irregularities, pregnancy, diabetes mellitus, thyroid conditions, recent COVID-19 infection, alterations in taste or smell, and medications affecting blood pressure. 23 participants were recruited and 7 participants became ineligible due to a variety of factors including: starting hormonal contraception, an irregular or missed cycle, <100 ng/mL E3G throughout periovulation, a lack of increased E3G at ovulation as compared to menstruation or lost to follow up. The participants in the control group consisted of 7 healthy, non-obese males between the ages of 18-26 years old.

Ovulation Tracking: Participants were asked to test their urine at the first urination of the day with Mira fertility MAX wands (San Francisco, CA) according to product instructions for 5 days prior to expected ovulation. Mira fertility MAX wands detect urine luteinizing hormone (LH), oestrone-3-glucuronide (E3G), and pregnanediol (PdG). E3G is a metabolite of estrone and is a marker of plasma 17-beta-estradiol. When participants' E3Gs rose above their menstruation baseline and reached > 100 ng/mL, they were asked to undergo the taste testing.

Biological males were also tested under the same conditions at comparable time differences (approximately 2 weeks apart) as a control for variation in taste testing.

Detection Threshold Testing: Participants underwent detection threshold testing with 1/8 log step serial dilutions of D-(+)-glucose (> 99.5%, Sigma-Aldrich, USA), sucralose and methyl-D-glucopyranoside (Sigma-Aldrich, USA). The participants were randomly presented with glucose or sucralose detection testing, followed by MDG detection testing. Detection threshold testing followed a 2-alternative-forced choice (2AFC) paradigm. Two medicine cups of Millipore water and dilute stimulus were presented to the participant in random order and the participant was asked which stimulus was "not water." A 4-down-1-up modified staircase method was used to obtain the oral detection threshold of the sweet stimulus. In this method, the participant is required to make the correct choice four times until the next more dilute stimulus is presented, and if the participant is wrong once, a more concentrated stimulus is presented in the next trial. Once the participant has made 5 reversals, the last 4 concentrations are averaged and defined as the detection threshold concentration for that stimulus. Participants wore nose clips throughout their testing.

Hedonic Rating Testing: Participants were trained to use the hedonic labeled magnitude scale. Participants were presented with three rows of randomized 450 mM and 900 mM glucose solutions and asked to taste and expectorate each solution and then rate their liking of the solution on a hedonic labeled magnitude scale. The solutions were presented in random order with a 30 second rinse of Millipore water in between each stimulus. Between each row there was a 2 minute break. Subjects did not wear nose clips for this part of the study.

ELIGIBILITY:
Inclusion Criteria:

* regular menstrual cycle of 21-35 days

Exclusion Criteria:

* hormonal contraceptives or other hormonal treatments
* a history of polycystic ovarian syndrome (PCOS)
* menstrual irregularities
* pregnancy
* diabetes mellitus
* thyroid conditions
* recent COVID-19 infection
* alterations in taste or smell
* medications affecting blood pressure

Ages: 18 Years to 46 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants were selected from residents in the general area around New Brunswick NJ where Rutgers University is located. Women and men were recruited of all available races and ethnicities.
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Oral Glucose Detection Threshold | Women were tested twice over the course of a cycle at menstruation and ovulation, and this was repeated for two cycles (across two months).
  Participants had an oral glucose detection threshold measured at menstruation (estrogen nadir) and peri-ovulation (estrogen peak). Men were tested twice two weeks apart over the same time frame as women.
Oral Sucralose Detection Threshold | Women were tested twice over the course of a cycle at menstruation and ovulation, and this was repeated for two cycles (across two months).
  Participants had an oral sucralose detection threshold measured at menstruation (estrogen nadir) and peri-ovulation (estrogen peak).
Oral MDG Detection Threshold | Women were tested twice over the course of a cycle at menstruation and ovulation, and this was repeated for two cycles (across two months).
  Participants had an oral s detect MDG (methyl-D-glucopyranoside) on threshold measured at menstruation (estrogen nadir) and peri-ovulation (estrogen peak).

SECONDARY OUTCOMES:
Concentrated Glucose Solution Preference | Women were tested twice over the course of a cycle at menstruation and ovulation, and this was repeated for two cycles (across two months).
  Participants tasted 450 and 900 mM glucose and rated liking on a labeled hedonic scale at menstruation (estrogen nadir) and peri-ovulation (estrogen peak).

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Breslin, PhD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Department of Nutritional Sciences, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
When published the data will be available upon request of the article contact.
Supporting Information: Study Protocol, SAP
Time Frame: March 2025 - February 2032
Access Criteria: Those requiring data for further analysis or for publication purposes at an institute of research or higher education may request information. Requests must describe the types of analyses that will be conducted.
URL: https://nutrition.rutgers.edu/faculty/paul-breslin.html